CLINICAL TRIAL: NCT02396381
Title: A Randomized, Controlled, 2-arm Parallel Group, Multi-center Study, to Evaluate Biological and Functional Changes in Healthy Smokers Switching to Tobacco Heating System 2.2 (THS 2.2) Compared to Continuing Smoking Conventional Cigarettes for 26 Weeks in an Ambulatory Setting
Brief Title: Evaluation of Biological and Functional Changes in Healthy Smokers After Switching to THS 2.2 for 26 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRHR-ERS-09-US; ZRHR-ERS-09-US (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Smoking
Keywords: Candidate modified risk tobacco product; Conventional cigarette; Exposure response; Smoking; Tobacco Heating System
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THS 2.2 (Experimental): Ad libitum use of THS 2.2
  Interventions: Other: THS 2.2
- CC (Active Comparator): Ad libitum use of CC
  Interventions: Other: CC

INTERVENTIONS:
Other: THS 2.2 — Ad libitum use of THS 2.2 in an ambulatory setting for 26 weeks
  Arms: THS 2.2
Other: CC — Ad libitum use of CC in an ambulatory setting for 26 weeks
  Arms: CC

SUMMARY:
The aim of the study is to demonstrate clinical, biological and functional health changes in smokers switching to the candidate modified risk tobacco product: Tobacco Heating System 2.2 (THS 2.2) as compared to smokers continuing smoking their conventional cigarettes (CC) over a 26-week period.

To characterize the study as successful, at least 5 clinical risk endpoints should move in the direction of smoking cessation and these results would be statistically significant. The main analysis will be defined a priori (using the Hailperin-Ruger approach) and will be made between THS 2.2 use and CC use as "per actual product used" and product use categories.

DETAILED DESCRIPTION:
The clinical, biological and functional endpoints to be measured in this study ("smoker's health profile") may characterize the modification of risk of smoking-related diseases.

Clinical risk endpoint to be assessed are selected based on a) their association to smoking-related diseases b) their association to smoking status, c) their reversibility upon smoking cessation, and d) their suitability to be measured with valid and robust methods in clinical studies.

The biological markers, functional markers and biomarkers of exposure (BoExp) with the strongest scientific evidence will constitute the 'smoker's health profile' and will be measured as the primary objective of the study.

Additional endpoints involved in the mechanistic of smoking-related diseases will be studied to provide additional scientific evidence to strengthen the primary objective.

The study will provide a perspective of product usage in a "real world setting" where smoking CC in addition to THS 2.2 may be expected.

ELIGIBILITY:
Inclusion Criteria:

* Current healthy smoker as judged by the Principal Investigator(s) or designee(s)
* Minimum age: 30 years old
* Have smoked for the last 10 years
* Have smoked more than 10 non menthol CC/day on average (no brand restriction) over the past year

Exclusion Criteria:

* Clinically relevant medical conditions that in the opinion of the investigators would jeopardize the safety of the participant.
* Subject who has (FEV1/FVC) < 0.7 and FEV1 < 80% predicted value at post-bronchodilator spirometry
* Subject with asthma condition (post-bronchodilator FEV1/FVC < 0.75 and reversibility in FEV1 ≥ 12% and > 200 mL from pre- to post-bronchodilator values)
* Subject who took or is taking concomitant medication which may have an impact on the "smoker's heath profile"
* Female subject is pregnant or breast feeding.
* Female subject who does not agree to use an acceptable method of effective contraception.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1039 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Danielle Armas, MD, Principal Investigator — Celerion Arizona; Leonard Dunn, MD, Principal Investigator — Clinical Research West Florida; Hugh Coleman, MD, Principal Investigator — Covance; George Stoica, MD, Principal Investigator — Compass Research; Mark Adams, MD, Principal Investigator — Central Kentucky Research Associate; Peter Davidson, MD, Principal Investigator — Celerion Lincoln; John Rubino, MD, Principal Investigator — PMG Research of Raleigh; George Raad, MD, Principal Investigator — PMG Research of Charlotte; Kevin Cannon, MD, Principal Investigator — PMG Research of Wilmington; Derek Schroder, MD, Principal Investigator — PMG Research of Cary; Stephanie Powell, MD, Principal Investigator — PMG Research of Bristol; William Smith, MD, Principal Investigator — NOCCR; Darrell Herrington, MD, Principal Investigator — Benchmark; Laurence Chu, MD, Principal Investigator — Benchmark; William Seger, MD, Principal Investigator — Benchmark; Lon Lynn, MD, Principal Investigator — Clinical Research West Florida; David Subich, MD, Principal Investigator — Compass Research; Isabel Kuhare-Arcure, MD, Principal Investigator — Midwest Clinical Research; Keith Scott, MD, Principal Investigator — National Clinical Research
Locations (19):
- United States (19):
  - Celerion Arizona, Tempe, Arizona
  - Clinical Research West Florida, Clearwater, Florida
  - Covance, Inc, Daytona Beach, Florida
  - Compass Research, Orlando, Florida
  - Clinical Research West Florida, Tampa, Florida
  - Compass Research, The Villages, Florida
  - Central Kentucky Research Associate, Lexington, Kentucky
  - Celerion Lincoln, Lincoln, Nebraska
  - PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - PMG Research of Bristol, Bristol, Tennessee
  - NOCCR, Knoxville, Tennessee
  - Benchmark, Austin, Texas
  - Benchmark, Fort Worth, Texas
  - Benchmark, San Angelo, Texas
  - National Clinical Research, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ludicke F, Ansari SM, Lama N, Blanc N, Bosilkovska M, Donelli A, Picavet P, Baker G, Haziza C, Peitsch M, Weitkunat R. Effects of Switching to a Heat-Not-Burn Tobacco Product on Biologically Relevant Biomarkers to Assess a Candidate Modified Risk Tobacco Product: A Randomized Trial. Cancer Epidemiol Biomarkers Prev. 2019 Nov;28(11):1934-1943. doi: 10.1158/1055-9965.EPI-18-0915. Epub 2019 Jul 3. PMID 31270101
- [Derived] Ansari SM, Lama N, Blanc N, Bosilkovska M, Donelli A, Picavet P, Baker G, Haziza C, Ludicke F. Evaluation of Biological and Functional Changes in Healthy Smokers Switching to the Tobacco Heating System 2.2 Versus Continued Tobacco Smoking: Protocol for a Randomized, Controlled, Multicenter Study. JMIR Res Protoc. 2018 Aug 24;7(8):e11294. doi: 10.2196/11294. PMID 30143474

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following randomization of 984 subjects, from 1039 enrolled subjects, one clinical site was terminated from this study due to non-GCP compliance.
  The safety population of 1012 subjects included all enrolled subjects except 27 subjects from the terminated site.
Groups:
- THS 2.2 Group: Randomized to Ad libitum use of THS 2.2 in an ambulatory setting for 26 weeks
- CC Group: Randomized to Ad libitum use of CC in an ambulatory setting for 26 weeks
Period: Overall Study
Arm/Group | THS 2.2 Group | CC Group
Started (Randomized) | 488 | 496
Full Analysis Set - As Exposed (FAS-EX) (Subjects with at least one record of reported use post-randomization.) | 414 | 443
Completed | 381 | 422
Not Completed | 107 | 74
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 33 | 24
Not completed — Lost to Follow-up | 49 | 31
Not completed — Protocol Violation | 1 | 0
Not completed — Site terminated by sponsor | 7 | 8
Not completed — Physician Decision | 5 | 5
Not completed — Pregnancy | 2 | 0
Not completed — Non-compliance with study procedures | 1 | 0
Not completed — Moved out of town/state | 1 | 3
Not completed — Could not complete visit | 1 | 0
Not completed — Possible conflict of interest | 1 | 0
Not completed — Randomization/Screening Error | 3 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - As Exposed (FAS-EX)
Groups:
- THS 2.2 Use: ≥1 THS 2.2 or CC, and ≥70% THS 2.2 use over the analysis period, and ≥70% THS 2.2 use on >50% of days in the analysis period.
- CC Use: ≥1 THS 2.2 or CC use, and <1% THS 2.2 use over the entire analysis period and <1% THS 2.2 use on ≥ 50% of days in the analysis period.
- Dual Use: ≥ 1 THS 2.2 or CC and, 1% ≤THS 2.2 <70% over the analysis period, or THS 2.2-use and CC-use categories do not apply to 50% of these days.
- Other Use: Subjects with missing product use data, subjects using e-cigarettes or other tobacco products, quitters, or subjects who switched across different use patterns between consecutive analysis periods.
- Total: Total of all reporting groups
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use | Total
Number analyzed (Participants) | 245 | 428 | 142 | 42 | 857
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (9.64) | 45.2 (9.55) | 43.8 (9.77) | 44.2 (8.14) | 44.6 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 182 | 63 | 14 | 353
  Male | 151 | 246 | 79 | 28 | 504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 28 | 7 | 1 | 53
  Not Hispanic or Latino | 228 | 400 | 135 | 41 | 804
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 0 | 6
  Asian | 2 | 5 | 0 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 0 | 3
  Black or African American | 42 | 74 | 25 | 10 | 151
  White | 195 | 341 | 113 | 30 | 679
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 2 | 1 | 10
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.9 (3.99) | 27.1 (4.13) | 26.9 (4.35) | 26.9 (5.12) | 27.0 (4.18)

OUTCOME MEASURES:

1. Primary Outcome: Levels of High Density Lipoprotein C (HDL-C).
Description: Concentrations measured in serum.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
mg/dL | 54.1 [51.4 to 56.7] | 50.9 [49.4 to 52.4] | 56.3 [52.7 to 59.9] | 52.8 [47.4 to 58.1]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will test if the mean level of HDL-C for THS-use is greater than for CC-use. The following hypothesis will be evaluated: H0: XTHS - XCC ≤ 0.0 HA: XTHS - XCC > 0.0 where XTHS and XCC are the adjusted means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Other; p < 0.001, Hailperin-Rüger; p-value less than 1.5625% would be considered statistically significant, following test multiplicity adjustment using the Hailperin-Rüger approach; LS Mean Difference = 3.09, 96.875% CI 2-sided [1.10 to 5.09]

2. Primary Outcome: Levels of White Blood Cells (WBC).
Description: Concentrations measured in blood.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: GI/L
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
GI/L | 6.98 [6.70 to 7.25] | 7.48 [7.28 to 7.69] | 7.41 [7.00 to 7.82] | 8.71 [7.80 to 9.62]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will test if the mean level of WBC for THS-use is lower than for CC-use. The following hypothesis will be evaluated: H0: XTHS - XCC ≥ 0.0 HA: XTHS - XCC < 0.0 where XTHS and XCC are the adjusted means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p = 0.001, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.420, 96.875% CI 2-sided [-0.717 to -0.123]

3. Primary Outcome: Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1).
Description: FEV1 post-bronchodilator and expressed as percentage predicted (FEV1 %pred).
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of predicted FEV1
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
Percent of predicted FEV1 | 95.4 [93.7 to 97.1] | 93.4 [92.0 to 94.8] | 93.7 [91.3 to 96.0] | 94.3 [89.3 to 99.4]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will test if the mean level of FEV1 for THS-use is greater than for CC-use. The following hypothesis will be evaluated: H0: XTHS - XCC ≤ 0.0 HA: XTHS - XCC > 0.0 where XTHS and XCC are the adjusted means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p = 0.008, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.28, 96.875% CI 2-sided [0.145 to 2.42]

4. Primary Outcome: Concentrations of Soluble Intercellular Adhesion Molecule 1 (sICAM-1).
Description: Concentrations measured in serum.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
ng/mL | 252 [239 to 266] | 266 [253 to 279] | 270 [253 to 288] | 273 [234 to 317]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis of sICAM-1 will test if the mean level of this clinical risk endpoint for THS-use is lower relative to CC-use. The following hypothesis will be evaluated: H0: XTHS / XCC ≥ 1.0 HA: XTHS / XCC < 1.0 where XTHS and XCC are the adjusted geometrical means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p = 0.030, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; % Reduction = 2.86, 96.875% CI 2-sided [-0.426 to 6.04] — Derived as 1 - LS Mean Ratio (THS / CC)

5. Primary Outcome: Concentrations of 11-dehydrothromboxane B2 (11-DTXB2).
Description: Concentrations measured in urine and expressed as concentration adjusted for creatinine.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
pg/mg creat | 496 [446 to 551] | 523 [482 to 568] | 532 [464 to 610] | 626 [504 to 777]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis of 11-DTX-B2 will test if the mean level of this clinical risk endpoint for THS-use is lower relative to CC-use. The following hypothesis will be evaluated: H0: XTHS / XCC ≥ 1.0 HA: XTHS / XCC < 1.0 where XTHS and XCC are the adjusted geometrical means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p = 0.193, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; % Reduction = 4.74, 96.875% CI 2-sided [-7.5 to 15.6] — Derived as 1 - LS Mean Ratio (THS / CC)

6. Primary Outcome: Concentrations of 8-epi-prostaglandin F2α (8-epi-PGF2α).
Description: as for outcome 5
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
pg/mg creat | 321 [299 to 344] | 351 [334 to 369] | 347 [318 to 377] | 335 [281 to 400]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis of 8-epi-PGF2α will test if the mean level of this clinical risk endpoint for THS-use is lower relative to CC-use. The following hypothesis will be evaluated: H0: XTHS / XCC ≥ 1.0 HA: XTHS / XCC < 1.0 where XTHS and XCC are the adjusted geometrical means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p = 0.018, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; % Reduction = 6.80, 96.875% CI 2-sided [-0.216 to 13.3] — Derived as 1 - LS Mean Ratio (THS / CC)

7. Primary Outcome: Concentrations of Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL).
Description: as for outcome 5
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
pg/mg creat | 144 [118 to 175] | 282 [254 to 314] | 286 [244 to 334] | 342 [254 to 460]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis of Total NNAL will test if the mean level of this clinical risk endpoint for THS-use is lower relative to CC-use. The following hypothesis will be evaluated: H0: XTHS / XCC ≥ 1.0 HA: XTHS / XCC < 1.0 where XTHS and XCC are the adjusted geometrical means of THS-use and CC-use, respectively. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p < 0.001, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; % Reduction = 43.5, 96.875% CI 2-sided [33.7 to 51.9] — Derived as 1 - LS Mean Ratio (THS / CC)

8. Primary Outcome: Percent Change From Baseline of Carboxyhemoglobin (COHb)
Description: Carboxyhemoglobin (COHb) is assayed from whole blood.
  Geometric Least Squares means are provided as descriptive statistics. Expressed as % of saturation of hemoglobin.
Time Frame: 26 Weeks
Population: Full Analysis Set - As Exposed (FAS-EX)
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 245 | 428 | 142 | 42
percentage change from baseline | 2.84 [2.51 to 3.20] | 4.38 [4.16 to 4.61] | 4.23 [3.80 to 4.70] | 5.59 [4.87 to 6.41]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will test if the mean level of COHb for THS-use is lower relative to CC-use. The following hypothesis will be evaluated: H0: XTHS / XCC ≥ 1.0 HA: XTHS / XCC < 1.0 where XTHS and XCC are the adjusted geometrical means of THS-use and CC-use. H0 is rejected with a type I error α = 1.5625% (one-sided test); Test type: Superiority; p < 0.001, Hailperin-Rüger; [statistical method as in outcome 1, analysis 1]; % Reduction = 32.2, 96.875% CI 2-sided [24.5 to 39] — Derived as 1 - LS Mean Ratio (THS / CC)

ADVERSE EVENTS:
Time Frame: The entire study duration per subject was between 32 to 38 weeks, including a Screening period of up to 42 days prior to enrollment, a 6 to 10-day run-in period prior to randomization, followed by a 26 week randomized exposure period. The end of study for a subject was defined as the check-out or the date of early termination of the subject plus the 28 day Safety Follow-up period, unless the subject was lost to follow-up.
Groups:
- Product Test: Enrolled subjects who participated in a product test, but were not randomized.
Arm/Group | THS 2.2 Group | CC Group | Product Test
All-Cause Mortality (participants affected / at risk) | 2/477 | 0/483 | 0/52
Serious Adverse Events (participants affected / at risk) | 6/477 | 7/483 | 0/52
Other Adverse Events (participants affected / at risk) | 23/477 | 29/483 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Group (N=477) | CC Group (N=483) | Product Test (N=52)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute, with Urosepsis and Nephrolithiasis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Head injury with seizure (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood and bereavement (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Metastases to small intestine with anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Vertebral osteophyte with Cervical myelopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Group (N=477) | CC Group (N=483) | Product Test (N=52)
Upper respiratory tract infection (Infections and infestations) | 23 (26) | 29 (33) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.